CLINICAL TRIAL: NCT04175457
Title: The Acute Effects of E-cigarette Inhalation on Vascular Function, Microcirculation and Thrombosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Umeå University (Other)
Responsible Party: Principal Investigator, Magnus Lundbäck, MD, Associate Professor, Karolinska Institutet
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 2018/2721-31/1
Record Dates: First submitted 2019-09-11; First posted 2019-11-25 (Actual); Last update posted 2020-03-19 (Actual); Status verified 2020-03

CONDITIONS: E-cigarette Use; Microcirculation; Thrombosis; Vascular Function; Blood Markers; Microvesicles; NETs
MeSH Terms: conditions — Vaping; Thrombosis | interventions — Electronic Nicotine Delivery Systems

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- e-cigarette inhalation with nicotine (Experimental): inhalation of e-cigarette vapor with nicotine for 30 minutes.
  Interventions: Other: e-cigarette
- e-cigarette inhalation without nicotine (Active Comparator): inhalation of e-cigarette vapor without nicotine for 30 minutes.
  Interventions: Other: e-cigarette

INTERVENTIONS:
Other: e-cigarette — E-cigarette inhalation for 30 minutes using e-cigarette with and without nicotine

SUMMARY:
This is a human randomized controlled cross-over study where the effects of e-cigarette inhalation (with or without nicotine) on vascular function, microcirculation and thrombosis is assessed.

DETAILED DESCRIPTION:
Twenty-two healthy, female and male occasional smokers or snus users (age 18-55, 10 cigarettes per month, 10 pouches of snus per month) will be included. Research subjects are required to refrain from intake of alcohol and caffeine during at least 24 hours prior to the exposure. Tobacco usage (including Swedish moist snuff) or e-cigarette usage is not permitted within 7 days prior to exposure.

All subjects have to complete a normal health declaration.

In a randomized cross-over fashion, all subjects will inhale vapor (30 puffs for 30 minutes) from one electronic cigarette, eVic-Primo SE (Shenzhen Joyetech Co., Ltd., China). in a specially prepared room with adequate ventilation.

There are plenty e-liquid manufacturers and distributors on the market. Independent content analysis showed that nicotine variation across e-liquid batches is low and that the amount of nicotine as stated by the manufacturer often is correct. E- liquid without any flavourings (Valeo laboratories GmbH, Germany) without and with nicotine (19 mg/ml) will be used. Content analysis is free available on the manufacturers homepage (http://www.e-liquid-wholesale.com). A third-generation EC is used with settings (Temperature 230°C, Effect 32 W, Resistance 0,20 Ω).

Research subjects are required to refrain from intake of alcohol during at least 24 hours prior to the exposure sequences, as well as caffeine for 12 hours. The two occasions will be separated by at least one week. Subjects rest for 15 minutes preceding the exposure.

Following the initial 15 minute rest the measurements for various cardiovascular endpoints will be performed at baseline and up to two hours following both exposures. This will be done with the following methods:

Measurement of vascular function

Photopletysmography (PPG) Arterial stiffness is an independent measure of vascular damage and risk, and is best assessed with the gold-standard technique pulse-wave velocity (PWV). However this method is technically demanding requiring special equipment (like SphygmoCor) and educated study personell. Finger photoplethysmography, however, is potentially providing the same information as PWV, and is ideal for continous measurment of arterial stiffness.

pulse propagation time (PPT), the interval from the systolic to the diastolic peak of the pulse wave. PPT is an upcoming marker for arterial stiffness and vascular aging. At the same time ECG and heat sounds by a microphone will be recorded making the analysis easier to validate.

Microcirculation Iontophoresis and laser speckle contrast imaging (LSCI) Microcirculation is assessed by a non-invasive method where two substances (acetylcholine and nitroprusside) is applied in a small chamber (0,5 ml) on the surface of the skin. Changes in microcirculation is measured with laser Doppler. The method is completely harmless and pain free. An uncommon but plausible side effect is local temporary skin rash.

For every heart-beat a pressure wave is generated reaching even the most peripheral parts of the body. By measuring changes in light absorption it is possible to assess distensions (even very small) in the peripheral arteries and arterioles in the subcutaneous tissue, in for example the tip of the finger. Microcirculation can also be measured by laser speckle contrast imaging (LSCI) which is a non-invasive completely pain free method for assessing microcirculation of the skin.

Blood pressure A semi-automatic oscillometric sphygmomanometer will be used to measure blood pressure and heart rate.

Blood sampling Blood samples will be drawn into test tubes containing 1/10 0.129 M sodium citrate, EDTA and serum at baseline, at 0 hour, 1 hour and 2 hours after exposure. Plasma is later collected after centrifugation at 2 000g for 20 min in room temperature (RT) and then frozen at -70°C until analysis.

Measurement of thrombus formation (T-TAS) T-TAS® (Total Thrombus-formation Analysis System) is a means of assessing thrombus formation during variable flow conditions using a small blood sample.

Measurement of cotinine Levels of cotinine will be measured in serum using a commercial available ELISA technique.

Through direct microscopy of the capillaries of the nail bed of one of the fingers capillary blood flow can be assessed (capillary blood cell velocity, CBV, mm/s). This is a completely pain free and non-invasive method that takes about 15 minutes to perform.

Measurement of MV Plasma is thawed and centrifuged at 2000g for 20 minutes at RT. The supernatant is then re- centrifuged, at 13 000g for 2 minutes at RT. 20 μl of sample is incubated for 20 minutes in dark with phalloidin-Alexa-660 (Invitrogen, Paisley, UK), lactadherin-FITC (Haematologic Technologies, Vermont, USA), CD42a-PE (Platelet-MP (PMP), BD, Clone Alma-16), CD45- PC7 (Leukocyte-MV (LMV), Beckman Coulter, Dublin, Ireland) and CD144-APC (Endothelial-MV (EMV), AH diagnostics, Stockholm, SWE). PMVs are also labeled with CD154-PE (CD40L, abcam, Cambridge, UK) and EMVs with CD62E (E-selectin, Beckman Coulter, Dublin, Ireland). MVs are measured by flow cytometry on a Beckman Gallios instrument (CA, USA). The MV-gate is determined using Megamix beads (BioCytex, Marseille, France), which is a mix of beads of with diameters of 0.5 μm, 0.9 μm and 3.0 μm, respectively. MVs are defined as particles less than 1.0 μm in size, negative to phalloidin (in order to exclude cell membrane fragments) and positive to lactadherin. Conjugate isotype- matched immunoglobulin (IgG1-FITC, IgG1-PE, IgG1-APC and IgG1- PC7) with no reactivity against human antigens is used as a negative control to define the background noise of the cytometric analysis. The absolute number of MVs is calculated by means of the following formula: (MV counted x standard beads ⁄ L) ⁄ standard beads counted, (FlowCount, Beckman Coulter).

To determine whether MVs are released due to activation or apoptosis MVs are labeled with SYTO 13. SYTO 13 (Molecular Probes) is cell permeable and has a high fluorescent yield when bound to DNA or RNA. Our hypothesis is that MVs released from apoptotic cells express more DNA or RNA.

Pro-coagulant effect of MVs In vitro experiments are performed to investigate the influence of MVs on thrombin generation, and the relative contribution of the negatively charged surface provided by MVs. Briefly plasma samples are thawed and after the centrifugation steps described above we further centrifuge the samples (twice 21 000g in 45 min, RT) to obtain an MV enrich pellet. The pellet is then added to commercial plasma (Haemochrom, Diagnostica, Essen, Germany) with no addition of TF or phospholipids. Thrombin generation in plasma is determined by using the calibrated automated thrombogram (CAT) as originally described by Hemker et al. The calculated area under the curve represents the total amount of thrombin generated over time and is called the endogenous thrombin potential (ETP). Time to the start of thrombin generation (lag time), maximal concentration of thrombin generation (peak thrombin) and time to maximal thrombin generation (time to peak thrombin) is also assessed in CAT analysis.

ELIGIBILITY:
Inclusion Criteria:

* Normal health declaration

Exclusion Criteria:

* Any form of cardiovascular disease
* Any form of pulmonary disease like asthma or COPD
* Any form of systemic or chronic disorder like rheumatologic or metabolic diseases. - Symptoms of infection or inflammation within 4 weeks of the study
* Pregnancy

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2019-12-05 (Actual); Primary Completion 2020-01-27 (Actual); Study Completion 2020-01-27 (Actual)

PRIMARY OUTCOMES:
microcirculation | change from baseline and 1 hour following exposures
  Iontophoresis and laser speckle contrast imaging (LSCI), Measurement of capillary blood flow (Capiflow), GlycoCheck system
thrombosis (total thrombus formation analysis system) | change from baseline, 30 minutes and 2 hour following exposures
  T-TAS (area under the curve, flow pressure change)

SECONDARY OUTCOMES:
arterial stiffness | change from baseline up to 3 hours following exposures
  Photopletysmography (PPG), arteriographyTensioMed, Budapest, Hungary,Sphygmocor AtCor Medical, EndoPAT (Itamar)
Microvesicles | change from baseline, 30 minutes and 2 hour following exposures
  microvesicles of leukocyte, endothelial and platelet origin (MVs/microliter)
NETs(neutrophil extracellular traps) | change from baseline, 30 minutes and 2 hour following exposures
  blood levels of H3Cit using ELISA
capillary microscopy | change from baseline to 1 hour following exposures
  capillary blood cell velocity, CBV, mm/s

CONTACTS AND LOCATIONS:
Overall Officials: Erik Näslund, MD, Prof, Study Director — Karolinska Institutet, Danderyd Hospital
Locations (1):
- Institutionen för kliniska vetenskaper, Danderyds sjukhus, Danderyd, Stockholm County, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kabele M, Lyytinen G, Bosson JA, Hedman L, Antoniewicz L, Lundback M, Mobarrez F. Nicotine in E-cigarette aerosol may lead to pulmonary inflammation. Respir Med. 2025 Jun;242:108101. doi: 10.1016/j.rmed.2025.108101. Epub 2025 Apr 14. PMID 40239848
- [Derived] Lyytinen G, Brynedal A, Anesater E, Antoniewicz L, Blomberg A, Wallen H, Bosson JA, Hedman L, Mobarrez F, Tehrani S, Lundback M. Electronic Cigarette Vaping with Nicotine Causes Increased Thrombogenicity and Impaired Microvascular Function in Healthy Volunteers: A Randomised Clinical Trial. Cardiovasc Toxicol. 2023 Aug;23(7-8):255-264. doi: 10.1007/s12012-023-09802-9. Epub 2023 Aug 7. PMID 37548804